CLINICAL TRIAL: NCT01831986
Title: Addition of Both Pregnenolone and L-theanine to Ongoing Antipsychotic Treatment for Schizophrenia and Schizoaffective Disorders: an 8-week, Randomized, Double-blind, Placebo-controlled Multicenter Study
Brief Title: Pregnenolone and L-theanine Augmentation in the Treatment for Schizophrenia and Schizoaffective Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Sha'ar Menashe Mental Health Center (Other)
Collaborators: Tirat Carmel Mental Health Center (Other Government)
Responsible Party: Principal Investigator, Michael Ritsner, MD, PhD, Head, Acute Department, Sha'ar Menashe Mental Health Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13-9-10
Record Dates: First submitted 2010-12-14; First posted 2013-04-15 (Estimated); Last update posted 2013-12-05 (Estimated); Status verified 2013-12

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Schizophrenia; Schizoaffective disorder; Pregnenolone; L-Theanine; Augmentation
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Pregnenolone; theanine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pregnenolone + L-Theanine (Experimental): The 60 participating subjects will be randomized into 2 groups: 30 patients will receive PREG (50 mg/day) with L-theanine (400 mg/day) and 30 patients will receive a placebo, each for 8 weeks in a double-blind manner.
  Interventions: Dietary Supplement: Pregnenolone and L-Theanine
- Sugar caps. (Placebo Comparator): Placebo (4 caps/day)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Pregnenolone and L-Theanine — Pregnenolone (50 mg/day) with L-theanine (400 mg/day)
  Arms: Pregnenolone + L-Theanine
Other: Placebo — Caps
  Arms: Sugar caps.

SUMMARY:
Schizophrenia (SZ) and schizoaffective (SA) disorders are comprised of several debilitating symptoms. It was suggested that compounds with neuroprotective effects might be useful in the management of SZ/SA symptoms. Our previous clinical trials indicated significant beneficial effects for augmentations with two different neuroprotective agents: Pregnenolone and L-Theanine. Pregnenolone (PREG) is a neurosteroid, which displays multiple effects on the central nervous system. Our recent 8-week, randomized, double-blind trial among patients with chronic SZ/SA disorders, in which PREG versus placebo and DHEA was added to antipsychotics, yielded encouraging results: PREG augmentation demonstrated significant amelioration of positive symptoms, EPS, as well as an improvement in attention, and working memory performance of SZ/SA disorder patients (Ritsner et al 2010). L-Theanine is a unique amino acid present almost exclusively in the tea plant. It possesses neuroprotective, mood-enhancing, and relaxation activities. L-theanine augmentation to antipsychotic therapy can ameliorate positive, activation, and anxiety symptoms in SZ/SA disorder patients (grant # 06TGF-911, (Ritsner et al 2010). This proposed study would extend our prior research with Pregnenolone and L-theanine by combining both agents versus placebo. We hypothesized that addition of both these compounds to ongoing antipsychotics would significantly improve the clinical status of SZ/SA patients.

Methods: In an 8-week, randomized, double-blind placebo-controlled trial a combination of PREG (50 mg/day) with L-theanine (400 mg/day) versus placebo will be added to the stable ongoing antipsychotic treatment of 200 patients with schizophrenia or schizoaffective disorders. This trial will be conducted at five sites in Israel. Participants will be assessed at baseline and after 2, 4, 6 and 8 weeks of treatment. A battery of research instruments will be used for the assessment of psychopathology, side effects, general functioning and quality of life

DETAILED DESCRIPTION:
This is a two-year randomized placebo-controlled double-blind investigation of the augmentation of PREG with L-theanine in the management of patients with SZ/SA. The study will consist of two phases: a 2-week continued stability (lead in) phase and an 8-week double-blind treatment phase. In the lead-in phase, patients receiving antipsychotic medication will remain on their maintenance regimen for at least two weeks. Clinical stability is defined as two consecutive weekly CGI ratings with no change in score, and with no more than a 20% change in PANSS total score. The treatment phase will be 8-week parallel groups, placebo-controlled, double-blind trial of adjunctively administered PREG with L-theanine or placebo. Assignment to PREG with L-theanine or placebo will be on a random, stratified (i.e., FGAs/SGAs, inpatient/outpatient) basis. PREG (50 mg/day) with L-theanine (400 mg/day) and placebo will be administered in divided doses in the form of capsules. If a patient relapses during the treatment phase of the study, the patient will be removed from the study. All attempts will be made to obtain end-of-study ratings. If such measures cannot be obtained, four- and six-week data, if collected prior to relapse, will be informative. Patients who fulfill the entry criteria will enter the 8-week double-blind treatment phase of the study. Assignment to PREG with L-theanine or placebo will be on a random, stratified (i.e., conventional/new generation antipsychotic treatment, inpatient/outpatient) basis. PREG (50 mg/day) with L-theanine (400 mg/day)/placebo will be administered in divided doses in the form of white capsules. If a patient relapses during the treatment phase of the study, the patient will be removed from the study. All attempts will be made to obtain end-of-study ratings. If such measures cannot be obtained, four- and eight-week data, if collected prior to relapse, will be informative.

Subjects will be assessed at baseline and after 2, 4, 6, and 8 weeks of treatment using psychiatric rating scales, and self-report questionnaires. Neurobiological (plasma cortisol, PREG, dehydroepiandrosterone, BDNF and other biologically active molecules) and immunological (the pro-inflammatory cytokines and others) testing will be conducted at baseline, and after treatment. The efficacy and safety of augmenting antipsychotic treatment of PREG with L-theanine will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-50 years, men or women.
* DSM-IV criteria for schizophrenia or schizoaffective disorder (American Psychiatric Association 2000).
* Subjects entering the study must score at least 4 on the Clinical Global Impression Scale (CGI-S).
* At least two weeks of ongoing treatment with current antipsychotic agents.
* No change in anticholinergic, or benzodiazepine medications for the pre-treatment stabilization period.
* Stable symptoms throughout the 2 week pre-treatment stabilization period.
* Ability and willingness to sign an informed consent form for participation in the study.

Exclusion Criteria:

* Evidence of serious neurologic or endocrine disorder, for example severe head trauma, seizure disorder, dementia, Cushings disease, or thyroid disorder, mental retardation, alcohol or drug abuse, substance dependence (other than nicotine dependence), or presenting symptoms likely substance-induced, as judged by a study physician.
* Unstable medical illness or neurologic illness (seizures, CVA); breast, uterine, or ovarian cancer.
* Patients with impaired renal function or with a history of significant impaired renal function will be excluded.
* Patients with significant suicidal risk will be excluded.
* Pregnant women, use of oral contraceptives or other hormonal supplementation such as estrogen. [Female patients will also have a pregnancy test.].
* Known allergy to study medication.
* Patients receiving mood-stabilizing medications.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-01; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
The Positive and Negative Syndrome Scale | 2 weeks

SECONDARY OUTCOMES:
Extrapyramidal Symptom Rating Scale | 2 weeks
Barnes Akathisia Scale | 2 weeks
The Liverpool University Neuroleptic Side Effect Rating Scale | 4 weeks
Global Assessment of Functioning | 4 weeks
Subjective Scale to Investigate Cognition in Schizophrenia | 4 weeks
Quality of Life Enjoyment and Satisfaction Questionnaire - Abbreviated version (Q-LES-Q-18) | 4 weeks
SANS | 2 weeks
Hamilton Anxiety Scale | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Ritsner, MD, PhD, Principal Investigator — Shaar Menashe MHC

REFERENCES:
- [Background] Ritsner MS, Gibel A, Shleifer T, Boguslavsky I, Zayed A, Maayan R, Weizman A, Lerner V. Pregnenolone and dehydroepiandrosterone as an adjunctive treatment in schizophrenia and schizoaffective disorder: an 8-week, double-blind, randomized, controlled, 2-center, parallel-group trial. J Clin Psychiatry. 2010 Oct;71(10):1351-62. doi: 10.4088/JCP.09m05031yel. Epub 2010 Jun 15. PMID 20584515
- [Background] Ritsner MS. Pregnenolone, dehydroepiandrosterone, and schizophrenia: alterations and clinical trials. CNS Neurosci Ther. 2010 Spring;16(1):32-44. doi: 10.1111/j.1755-5949.2009.00118.x. PMID 20070787
- [Background] Ritsner M, Maayan R, Gibel A, Weizman A. Differences in blood pregnenolone and dehydroepiandrosterone levels between schizophrenia patients and healthy subjects. Eur Neuropsychopharmacol. 2007 Apr;17(5):358-65. doi: 10.1016/j.euroneuro.2006.10.001. Epub 2006 Nov 21. PMID 17123790
- [Derived] Kardashev A, Ratner Y, Ritsner MS. Add-On Pregnenolone with L-Theanine to Antipsychotic Therapy Relieves Negative and Anxiety Symptoms of Schizophrenia: An 8-Week, Randomized, Double-Blind, Placebo-Controlled Trial. Clin Schizophr Relat Psychoses. 2018 Spring;12(1):31-41. Epub 2015 Jul 28. PMID 26218236